CLINICAL TRIAL: NCT04534920
Title: Comparison of Sample Characteristics Between the Subjects Who Received Strattice Mesh for Abdominal Wall Reconstruction at Westchester Medical Center vs Americas Hernia Society Quality Collaborative (AHSQC) Registry Dataset
Brief Title: Comparison of Sample Characteristics Between Subjects Who Received Strattice Mesh for Abdominal Wall Reconstruction
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: New York Medical College (Other)
Responsible Party: Principal Investigator, Rifat Latifi, The Felicien Steichen Professor and Chairman of Surgery, New York Medical College
Other Study IDs: 14073
Record Dates: First submitted 2020-08-25; First posted 2020-09-01 (Actual); Last update posted 2021-09-01 (Actual); Status verified 2021-08

CONDITIONS: Hernia
MeSH Terms: conditions — Hernia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Two different datasets from Institutional Review Board (IRB) approved studies L#12,083 and L#12,086 will be used to compare the sample characteristics between subjects who received Strattice mesh for abdominal wall reconstruction at Westchester Medical Center and Americas Hernia Society Quality Collaborative (AHSQC) registry.

DETAILED DESCRIPTION:
Abdominal wall defects or hernias are commonly seen after open surgery performed electively or under emergent conditions. During the last decade numerous advances have been made in the management of patients with abdominal wall defects. These defects are repaired by various surgical techniques including mesh repair (synthetic vs. biologic), primary repair, etc. However, the outcomes of patients after these injuries are highly variable and many of these patients suffer from in-hospital complications, mesh infections requiring explantation, and recurrence. Various factors play a role in the final outcome of the patient. These include factors associated with the reasons for initial surgery or disease (trauma or emergency general surgery), patient demographics (age, gender, co-morbidities), preoperative features (hemoglobin and other biochemical indicators, surgical technique used during the repair and use of repair (onlay, inlay, retro rectus) and the types of mesh used.

Study Design Two different datasets from Institutional Review Board (IRB) approved studies L#12,083 and L#12,086 will be used to compare the sample characteristics between subjects who received Strattice mesh for abdominal wall reconstruction at Westchester Medical Center and Americas Hernia Society Quality Collaborative (AHSQC) registry.

Primary Objective: To determine the degree to which our sample of Strattice® recipients resemble AHSQC Strattice® recipients.

Study Summary:

This study involves two different datasets from our existing studies L#12083 and L#12,086 which are approved by New York Medical College, IRB on 6/14/2017and 7/7/2017 respectively.

Study L#12,083 is a retrospective data collection of subjects who had abdominal wall reconstruction and received Strattice mesh during 1/1/2011 to 12/31/2018 at Westchester Medical Center. A total of 105 records from this study will be used for comparison study. Study L#12086 is a prospective study of subjects who had abdominal wall reconstruction using biological mesh. A total of 77 records will be used from this study. From both the studies combined we have about a total of 182 records of extracted data and same data variables will be used to compare with AHSQC registry. The data that will be compared includes preoperative info, hospital course, complications, re-hospitalizations and 2weeks follow-up.

Research Subject Population:

Number of Subjects Total of 182 records met the inclusion criteria and data has been collected.

Gender of Subjects There will be no gender based restrictions for this study.

Age of Subjects Subjects 18 to 85 years old will be included in this study.

ELIGIBILITY:
Inclusion Criteria:

* Subjects 18 to 85 years old
* Subjects who had complex abdominal wall reconstruction and received biologic mesh are included in the study

Exclusion Criteria:

* Subjects below 18 years of age and above the age of 85 years are excluded.
* Any hernia repair not using biologic mesh are excluded.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All male and female subjects who were between 18 to 85 years old, who had complex abdominal wall reconstruction at Westchester Medical Center and received biologic mesh during 1/1/2011 to 12/31/2018 are included in this study.
Sampling Method: Probability Sample
Enrollment: 182 (Actual)
Dates: Start 2020-07-27 (Actual); Primary Completion 2021-12-13 (Estimated); Study Completion 2021-12-13 (Estimated)

PRIMARY OUTCOMES:
comparison of sample characteristics between WMC Strattice® recipients and AHSQC Strattice® recipients | from 1/1/2011 to 12/31/2018
  Comorbidities, operative details, mesh size and location, number of drains, surgical site infection and readmissions.

CONTACTS AND LOCATIONS:
Overall Officials: Rifat Latifi, MD, Principal Investigator — Chairman Department of Surgery
Locations (1):
- Westchester Medical center, Valhalla, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided
no plan